CLINICAL TRIAL: NCT03316443
Title: A Prospective Randomized Comparative Study of Glidescope Versus Macintosh Laryngoscope in Adult Hypertensive Patients
Brief Title: A Comparative Study of Glidescope Versus Macintosh Laryngoscope in Adult Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Mahmoud Othman, professor of Anesthesia and surgical ICU, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MS/17.10.93
Record Dates: First submitted 2017-10-12; First posted 2017-10-20 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Hypertensive Patients
Keywords: Glidescope,Macintosh, Laryngscope, intubation,Hypertension.

STUDY DESIGN:
Intervention Model Description: Eligible 90 adult patients will be randomly allocated by a computer-generated randomization sequence into 2 equal groups:
  Macintosh group: 45 patients will be intubated by Macintosh laryngoscope (Group M).
  Glidescope group: 45 patients will be intubated by Glidescope (Group G).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group G) (Active Comparator): Glidescope group: 45 patients will be intubated by Glidescope (Group G). For endotracheal intubation with glidoscope, size 3 blade will be used in all of the cases. Glidoscope will be advanced gently in the oral cavity (in the midline) and walked down the tongue. The scope will be further advanced into the vallecula and gentle lifting force will be applied for visualization of the glottis. Endotracheal tube will be loaded on specific rigid stylet with 60 degree bent and will be advanced into the trachea by the same operator.
  Interventions: Device: Glidescope
- (Group M) (Experimental): Macintosh group: 45 patients will be intubated by Macintosh laryngoscope (Group M).The patient will be intubated by suitable sized tube (in males 8 mm and in females 7.5 mm internal diameter). In Macintosh group we will use a blade size 3 at first, the laryngoscope will be advanced in patient mouth displacing the tongue laterally till the laryngoscope reach the vallecula and then gentle lifting will be applied till visualization of the laryngeal inlet then the tube will be advanced
  Interventions: Device: Macintosh

INTERVENTIONS:
Device: Glidescope — The patient will be intubated by suitable sized tube (in males 8 mm and in females 7.5 mm internal diameter).
  For endotracheal intubation with glidescope, size 3 blade will be used in all of the cases. Glidoscope will be advanced gently in the oral cavity (in the midline) and walked down the tongue. The scope will be further advanced into the vallecula and gentle lifting force will be applied for visualization of the glottis. Endotracheal tube will be loaded on specific rigid stylet with 60 degree bent and will be advanced into the trachea by the same operator.
  Systolic, diastolic, mean arterial blood pressure and heart rate will be recorded at the following time points: T1: before anesthesia, T2: after induction and immediately before intubation, T3: immediate after completion of intubation, T4: after 1 minute of intubation, T5: after 2 minutes of intubation, T6: after 3 minutes of intubation, T7: after 5 minutes of intubation, T8: after 10 minutes of intubation.
  Arms: (Group G)
Device: Macintosh — The patient will be intubated by suitable sized tube (in males 8 mm and in females 7.5 mm internal diameter). In Macintosh group we will use a blade size 3 at first. The laryngoscope will be advanced in patient mouth displacing the tongue laterally till the laryngoscope reach the vallecula and then gentle lifting will be applied till visualization of the laryngeal inlet then the tube will be advanced.Systolic, diastolic, mean arterial blood pressure and heart rate will be recorded at the following time points: T1: before anesthesia, T2: after induction and immediately before intubation, T3: immediate after completion of intubation, T4: after 1 minute of intubation, T5: after 2 minutes of intubation, T6: after 3 minutes of intubation, T7: after 5 minutes of intubation, T8: after 10 minutes of intubation.Maximal arterial blood pressure and heart rate changes will be recorded
  Arms: (Group M)

SUMMARY:
Hemodynamic response to laryngoscopy and tracheal intubation remain of utmost concern in anesthesia practice. Sympathetic stimulation and adverse physiologic events could be tolerated by healthy individuals, but they may be detrimental in hypertensive patients.

The magnitude of hemodynamic response of intubation is related to the degree of manipulation of the oropharyngeo-laryngeal structures. Unlike Macintosh laryngoscope,Glidescope is a device that does not require alignment of oropharyngeal axis to visualize the glottis.It needs less upward lifting force with less manipulation of pharyngeal structures during the intubation.

It was reported that Glidescope had no significant advantage over Macintosh in attenuating circulatory response to endotracheal intubation in normotensive patients.Till now no clinical trials investigate the hemodynamic effects of Glidescope in hypertensive patients.The investigators hypothesized that the Glidescope will induce less hemodynamic changes among hypertensive patients during endotracheal intubation.So the study was designed to compare effects of Glidescope versus Macintosh laryngoscope in hypertensive patients with special regard to hemodynamics and intubation conditions.

DETAILED DESCRIPTION:
This is prospective randomized study will performed at Urology and Nephrology Centre, Mansoura University after approval from Institutional Research Board, Mansoura University.Patients were interviewed and written informed consent will be obtained from selected patients scheduled for different urological surgeries.

Eligible adult patients will be randomly allocated by a computer-generated randomization sequence into 2 equal groups:

Macintosh group: 45 patients will be intubated by Macintosh laryngoscope(Group M).

Glidescope group: 45 patients will be intubated by Glidescope(Group G).

Preoperative assessment:

All patients will be assessed preoperatively by:

1. History taking (for medical and surgical history)
2. Physical examination (including heart, blood pressure, electrocardiogram, chest auscultation and difficult airway assessment)
3. Laboratory investigation (complete blood picture, renal and liver function tests and bleeding profile).

The day before surgery, the study protocol will explained to all patients and the patients will fast for 6 hours before the surgery. All the patients will receive their antihypertensive medications till the morning of surgery

On arrival to the operation room:

Routine monitoring including: electrocardiogram, non-invasive blood pressure and pulse oximetry will be set, Peripheral intravenous cannula will be inserted and acetated Ringer will be started at rate of 4ml/kg/h.

Anesthetic management:

The induction will be similar in both groups; Pre-oxygenation for 5 minutes will be done in all patients and then they will receive 0.02 mg/Kg midazolam, 1μg/Kg fentanyl, 2mg/kg Propofol slowly until loss of verbal contact and rocurronium 0.6 mg/kg intravenously.Till the establishment of adequate neuromuscular block, the patients' ventilation will be assisted manually using a face mask. During this period the patients' lungs will be ventilated with 100% oxygen.

After establishment of adequate neuromuscular block after 3 minutes, the trachea will be intubated using either glidescope or Macintosh laryngoscope.The patient will be intubated by suitable sized tube (in males 8 mm and in females 7.5 mm internal diameter). In Macintosh group we will use a blade size 3, the laryngoscope will be advanced in patient mouth displacing the tongue laterally till the laryngoscope reach the vallecula and then gentle lifting will be applied till visualization of the laryngeal inlet then the tube will be advanced.For endotracheal intubation with glidescope, size 3 blade will be used in all of the cases. Glidescope will be advanced gently in the oral cavity (in the midline) and walked down the tongue. The scope will be further advanced into the vallecula and gentle lifting force will be applied for visualization of the glottis. Endotracheal tube will be loaded on specific rigid stylet with 60 degree bent and will be advanced into the trachea by the same operator.

External pressure to the front of the neck will be applied on request of the operator by another anesthetist.After placement of the endotracheal tube, the cuff of the tube will be inflated gradually with and the chest will be auscultated to ensure proper tracheal positioning and to exclude bronchial intubation and then the tube will be fixed.

All the intubations will be performed by a well-trained anesthetist. The intubation attempt failure will be defined when the intubation time exceed 120 seconds, esophageal intubation occurred or desaturation with arterial oxygen saturation dropped below 90%. Three attempts will only allow,then anesthesia will be carried out according to decision of the attending anesthetist with exclusion of the case from the study. Face-mask intermittent positive pressure ventilation will be carried out in-between the attempts.

The intubation condition will be assessed using first attempt success rate, number of attempts, intubation time and Cormack Lehane score. The intubation time is defined as the period from termination of face mask oxygenation till the appearance of carbon dioxide trace after positive pressure ventilation.

Cormack Lehane score is based on the laryngoscopic view as following: grade 1 full view of the glottis, grade 2 partial view of the glottis, grade 3 only the epiglottis appear and grade 4 neither the glottis nor the epiglottis appear

Monitoring:

Systolic, diastolic, mean arterial blood pressure and heart rate will be recorded at the following time points: T1: before anesthesia, T2: after induction and immediately before intubation, T3: immediate after completion of intubation, T4: after 1 minute of intubation, T5: after 2 minutes of intubation, T6: after 3 minutes of intubation, T7: after 5 minutes of intubation, T8: after 10 minutes of intubation.Maximal blood pressure and heart rate changes will be recorded

Postoperative follow up:

The patient will be assessed 24 hours postoperatively for the sore throat and hoarseness of voice according to the 4-point score

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 20 year old.
* Patients classified by the American society of anesthesiologist as 2 or 3 with controlled hypertension.
* Patients with body mass index less than 35.
* Mallampati score 1 or 2, thyromental distance more than 4 cm and central incisor interdistance more than 3 cm will included.

Exclusion Criteria:

* Patient refusal.
* Patient with uncontrolled hypertension (patients diagnosed as uncontrolled hypertension if they have history of hypertension and systolic blood pressure after 3 measures after admission exceeding 150 mmHg despite of regular antihypertensive therapy).
* Patient with major cardiac diseases (e.g cardiomyopathy).
* Patient with cerebrovascular accidents.
* Patient with history of difficult intubation.
* Patients at risk of aspiration who require rapid sequence induction.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Arterial blood pressure changes | During 10 minutes after endotracheal inubation.
  Systolic arterial blood pressure changes with the use of each device for endotracheal intubation.
Arterial blood pressure changes | During 10 minutes after endotracheal intubation.
  Diastolic arterial blood pressure changes with the use of each device for endotracheal intubation.
Arterial blood pressure changes | During 10 minutes of trial of endotracheal intubation.
  Mean arterial blood pressure changes with the use of each device for endotracheal intubation.
Heart rate changes | During 10 minutes of trial of endotracheal intubation.
  Heart rate changes with the use of each device for endotracheal intubation.

SECONDARY OUTCOMES:
Success rate of endotracheal intubation with each device. | During intraoperative trial of endotracheal intubation.
  First attempt success rate for endotracheal intubation completion.
Endotracheal intubation time with each device. | During intraoperative trials of endotracheal intubation.
  Total time needed from end of mask ventilation untill endotracheal intubation completion with appearance of CO2 traces.
Attempts of endotracheal intubation with each device. | During intraoperative trials of endotracheal intubation.
  Number of attempts needed for completion of endotracheal intubation.
severity of sore throat with each device. | 24 hours after endotracheal intubation
  Sore throat will be graded as none, mild (less severe than with common cold), moderate (similar to common cold) and severe (more severe than with common cold).
severity of hoarseness of voice with each device. | 24 hours after endotracheal intubation
  Hoarseness of voice will be graded as none, mild (noted only by the patient), moderate (obvious to the observer) and sever (like aphonia).

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M Othman, MD, Principal Investigator — Faculty of Medicine, Mansoura University.
Locations (1):
- Mansoura faculty of medicine, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided